CLINICAL TRIAL: NCT07104669
Title: Sports Nutrition Assessment Program at the University of Alicante
Brief Title: Sports Nutrition Assessment Program
Acronym: NutriEvalUA
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Jose Miguel Martinez Sanz, Associate Professor. Director of the Research Group on Applied Dietetics, Nutrition and Body Composition. Nursing Department. Faculty of Health Sciences. University of Alicante., University of Alicante
Other Study IDs: UA-2025-07-15
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Diet Habit; Body Weight; Athlete Foot
Keywords: sport nutrition; dietary-nutritional assessment; athletes; questionnaires
MeSH Terms: conditions — Feeding Behavior; Body Weight; Tinea Pedis | interventions — Diet; Exercise; Body Composition; Organism Hydration Status; Health Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- male: adults male athletes
  Interventions: Other: diet; Other: Physical activity; Other: body composition; Other: hydration status; Other: health status
- female: adults female athletes
  Interventions: Other: diet; Other: Physical activity; Other: body composition; Other: hydration status; Other: health status

INTERVENTIONS:
Other: diet — diet adherence
Other: Physical activity — Physical activity level
Other: body composition — body composition assessment
Other: hydration status — hydration status assessment
Other: health status — perception of health status

SUMMARY:
The NutriEvalUA program is an observational study aiming to assess the nutritional status, body composition, hydration, physical activity, and health indicators in university athletes. The main objective is to describe and evaluate dietary habits, supplement use, physical condition, and related risk factors to improve health and sports performance in this population. The main question it aims to answer is: What is the nutritional, body composition, hydration, physical activity, and general health profile of university athletes at the University of Alicante, and which factors are associated with potential risks to their performance and well-being?

DETAILED DESCRIPTION:
University athletes represent a population with specific nutritional and physiological needs. Despite their active lifestyle, there is often a lack of systematic evaluation protocols focused on their health and performance. NutriEvalUA addresses this gap through a comprehensive assessment protocol including anthropometry, body composition, dietary habits, physical activity levels, hydration status, and health-related questionnaires (e.g., sleep, disordered eating, exercise addiction).

This cohort study is carried out in collaboration with sports teams affiliated with the University of Alicante. The information obtained will help identify patterns, risks, and opportunities for nutritional intervention, supporting evidence-based strategies to optimize performance and promote long-term health.

ELIGIBILITY:
Inclusion Criteria:

* Acceptation of informed consent

Exclusion Criteria:

* No attendance to the evaluations
* Reporting less than 80% of assistance to physical activity sessions reported by trainer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University athletes who train and compete on the University of Alicante's sports teams
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Diet Adherence | 5 years
  Low, moderate or high

SECONDARY OUTCOMES:
Physical Activity Level | 5 years
  Low, moderate or high
Changes in Body Composition | 5 years
  Change in body composition (fat mass and muscle mass) by anthropometric evaluation
Hydration status | 5 years
  normohydrated, dehydrated, very dehydrated
perception of health status | 5 years
  very good, good, average, bad, very bad

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences. University of Alicante, San Vicent del Raspeig, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
The data are available from the authors on request from the IP JMMS (josemiguel.ms@ua.es).

REFERENCES:
- [Background] Lachat C, Hawwash D, Ocke MC, Berg C, Forsum E, Hornell A, Larsson C, Sonestedt E, Wirfalt E, Akesson A, Kolsteren P, Byrnes G, De Keyzer W, Van Camp J, Cade JE, Slimani N, Cevallos M, Egger M, Huybrechts I. Strengthening the Reporting of Observational Studies in Epidemiology-Nutritional Epidemiology (STROBE-nut): An Extension of the STROBE Statement. PLoS Med. 2016 Jun 7;13(6):e1002036. doi: 10.1371/journal.pmed.1002036. eCollection 2016 Jun. PMID 27270749
- [Background] Serafini S, Charrier D, Izzicupo P, Esparza-Ros F, Vaquero-Cristobal R, Petri C, Mecherques-Carini M, Baglietto N, Holway F, Tinsley G, Paoli A, Campa F. Anthropometric-based predictive equations developed with multi-component models for estimating body composition in athletes. Eur J Appl Physiol. 2025 Mar;125(3):595-610. doi: 10.1007/s00421-024-05672-3. Epub 2024 Dec 6. PMID 39641837
- [Background] Sebastia-Rico J, Soriano JM, Sanchis-Chorda J, Garcia-Fernandez AF, Lopez-Mateu P, de la Cruz Marcos S, Martinez-Sanz JM. Analysis of Fluid Balance and Urine Values in Elite Soccer Players: Impact of Different Environments, Playing Positions, Sexes, and Competitive Levels. Nutrients. 2024 Mar 21;16(6):903. doi: 10.3390/nu16060903. PMID 38542815
- [Background] Capling L, Beck KL, Gifford JA, Slater G, Flood VM, O'Connor H. Validity of Dietary Assessment in Athletes: A Systematic Review. Nutrients. 2017 Dec 2;9(12):1313. doi: 10.3390/nu9121313. PMID 29207495